CLINICAL TRIAL: NCT04877002
Title: Novel Salivary Rapid Testing of SARS_CoV_2
Brief Title: Performance Study of SONA Saliva C-19 Rapid Test
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited participants
Sponsor: Sona Nanotech Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT002-SalC19RT
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Sars-CoV-2 Infection; Corona Virus Infection
Keywords: Antigen; COVID19; Rapid Test; Saliva
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to validate the performance of the Sona Saliva C-19 rapid Test for rapid detection of SARS_CoV_2 infection when using saliva specimens. A prospective randomized and blinded study to evaluate a rapid point of care antigen test for the detection of viral proteins and compared against an approved RT-PCR test.
  Saliva samples will be collected along with the current standard of care collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS_CoV_2 Antigen Rapid Test (Experimental): The same group of patients participated in two arms of the study:
  One arm was for obtaining performance data of the Sona Saliva C-19 Rapid test and the comparator arm was to obtain data from the primary care route using approved RT-PCR testing.
  Interventions: Diagnostic Test: Sona Saliva C-19 Rapid Test

INTERVENTIONS:
Diagnostic Test: Sona Saliva C-19 Rapid Test — Rapid Antigen diagnostic device performance comparative to RT-PCR

SUMMARY:
The Sona Saliva C-19 Rapid Test is a bioassay intended for rapid point-of-care detection of the SARS-CoV-2 virus. Performance of the Sona Saliva C-19 Rapid Test assay will be assessed by comparison to a RT-PCR reference method

DETAILED DESCRIPTION:
The clinical performance of the Sona Saliva C-19 Rapid Test will be evaluated in a prospective clinical study conducted at a single (1) investigational site in Toronto, Cananda.

Consenting patients of ages 18+, any gender, or race/ethnicity who presents at the test site with COVID-19 like symptoms during the 2021 COVID-19 season will be asked to take part in the study, will be sequentially enrolled and tested.

Trained operators with laboratory experience who have received training on the use of the Sona Saliva C-19 Rapid Test will conduct the testing and represent the intended users.

A subject's participation in this study will consist of a single visit. Following the completion of the informed consent process, study questionnaire and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number, be asked to provide a sample for testing.

ELIGIBILITY:
Inclusion Criteria:

Up to 500 subjects will be screened, consented, and enrolled to obtain a minimum of 50 eligible candidates. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Presenting to the Emergency Department at HRH.
2. Receiving a COVID-19 RT-PCR test as per standard pathway of care.
3. Provide written informed consent.
4. Patients must be presenting or have experienced at least one (1) or more signs or symptoms of COVID-19 within ≤ 7 days:

   1. Fever as self-described or measured ≥ 38 °C (100.4°F)
   2. Chills
   3. Cough
   4. Shortness of breath
   5. Congestion or runny nose
   6. Difficulty Breathing
   7. Muscle or Body Aches
   8. Vomiting
   9. Diarrhea
   10. New loss of sense of taste or smell
   11. Headache
   12. General malaise
   13. Sore Throat

Exclusion Criteria:

1. Asymptomatic patients.
2. Patients unable to provide a saliva sample.
3. Patients unable to give consent.
4. Patients who will not be receiving a nasopharyngeal RT-PCR test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Percent Positive Agreement and Negative Percent Agreement | 35 days from last patient enrolment
  Calculate the performance of the Sona Saliva C-19 Rapid Test when compared to RT- PCR using nasopharyngeal swab specimens.

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobs, Dr, Principal Investigator — Humber River Hospital
Locations (1):
- Humber River Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No